CLINICAL TRIAL: NCT04716582
Title: The Effect of Different Ways of Sitting on Cognitive Performance and Muscle Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DSIT
Record Dates: First submitted 2020-09-21; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Sedentary Behavior; Light Intensity Physical Activity
Keywords: sedentary behavior; light physical activity; executive function; active sitting
MeSH Terms: conditions — Sedentary Behavior | interventions — Sitting Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SIT group (Experimental): participants will sitting 4 hours continuously.
  Interventions: Behavioral: uninterrupted sitting
- INTERRUPT group (Experimental): participants will sitting 25 minutes with 5 minutes walking per half hour,40minutes walking in total
  Interventions: Behavioral: Sitting interrupted by light physical activity
- COGN group (Experimental): participants will perform GED test as cognitive loading task during 4-hour sitting
  Interventions: Behavioral: Sitting with cognitive task

INTERVENTIONS:
Behavioral: Sitting interrupted by light physical activity — Each 30 minutes will be 25 minutes sitting followed by 5 minutes walking that designed as prescribed walking route outside laboratory corridor.
  Other Names: INTERRUPT
  Arms: INTERRUPT group
Behavioral: Sitting with cognitive task — Participants will perform online cognitive task during prolonged sitting.
  Other Names: COGN
  Arms: COGN group
Behavioral: uninterrupted sitting — Participants will watch documentary during prolonged sitting.
  Other Names: SIT
  Arms: SIT group

SUMMARY:
Academic educations concurs with a lot of sitting. Studies have shown that prolonged sitting not only has disruptive effects on physical health, but also influence mental health and cognition negatively. For physical health evidence grows that short light intense interruptions of sitting time effectively counterbalance the impact of prolonged sitting. It is not clear of light intense physical activity breaks have a similar positive effect on cognitive performance. Also, it is unclear whether cognitive loading might be able to compensate the impact of prolonged sitting.This study compares the effects of uninterrupted sitting with or without cognitive loading and interrupted sitting on cognitive functioning; muscle activation of leg and trunk muscles under various modes of sitting with walking, in order to calibrate the physical impact of different sitting modes.

DETAILED DESCRIPTION:
healthy university students will attend three separate intervention visits with 6-days (no more than 14 days) washout in between: 1) uninterrupted sitting (SIT); 2) uninterrupted sitting with a cognitive task (COGN); 3) sitting interrupted by light physical activity (INTERRUPT). For the SIT and INTERRUPT conditions, subjects watch a series of documentaries while sitting. In the COGN condition, while sitting, participants undergo the online GED test as cognitive load. Four cognitive tests (D2 test, stroop test, trail making test and 2-BACK test) and mood states will be performed before and after each intervention. On a separate day, using surface electromyography, activations of major leg and trunk muscles of sitting on chair, active and passive sitting on a yoga ball and walking were assessed.

ELIGIBILITY:
Inclusion Criteria:

* age 18-30 years
* BMI between 18-28
* steady dietary habits
* generally healthy
* Female on contraceptive pills/Male

Exclusion Criteria:

* High score (score: 11-21) in the Hospital Anxiety and Depression Scale

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive processes as assessed using Stroop test | change from baseline after 4 hour intervention on day1, day8, day16
  Stroop test is a computer-based Stroop word and color test, including congruent trials and incongruent trials to assess inhibition. Reaction time and accuracy of the Stroop test will be collected before and after the intervention
Cognitive processes as assessed using D2 attention test | change from baseline after 4 hour intervention on day1, day8, day16
  D2 attention test is a paper and pencil test to assess attention. Concentration performance will be collected before and after the intervention.
Cognitive processes as assessed using N back test | change from baseline after 4 hour intervention on day1, day8, day16
  N back test is a computer-based test, including target images and non-target images. this test is for updating and working memory. The correct reaction number of N back test will be collected before and after the intervention.
Cognitive processes as assessed using Trail making test | change from baseline after 4 hour intervention on day1, day8, day16
  Trail making test is a computer-based test to assess task-switching. reaction time and accuracy of the trail making test will be collected before and after the intervention.

SECONDARY OUTCOMES:
mood status assessed by tension score | change from baseline after 4 hour intervention on day1, day8, day16
  mood questionnaire(an abbreviated version of Profile of Mood States (POMS)) will be used before and after the intervention, such as tension, anger, depression, vigor, esteem-related effect, confusion, fatigue, total mood level data included. The scale is 0 to 4.
mood status assessed by anger score | change from baseline all mood outcomes after 4 hour intervention on day1, day8, day16
  mood questionnaire(an abbreviated version of Profile of Mood States (POMS)) will be used before and after the intervention, such as tension, anger, depression, vigor, esteem-related effect, confusion, fatigue, total mood level data included. The scale is 0 to 4.
mood status assessed by depression score | change from baseline all mood outcomes after 4 hour intervention on day1, day8, day16
  mood questionnaire(an abbreviated version of Profile of Mood States (POMS)) will be used before and after the intervention, such as tension, anger, depression, vigor, esteem-related effect, confusion, fatigue, total mood level data included. The scale is 0 to 4.
mood status assessed by vigor score | change from baseline all mood outcomes after 4 hour intervention on day1, day8, day16
  mood questionnaire(an abbreviated version of Profile of Mood States (POMS)) will be used before and after the intervention, such as tension, anger, depression, vigor, esteem-related effect, confusion, fatigue, total mood level data included. The scale is 0 to 4.
mood status assessed by esteem-related effect score | change from baseline all mood outcomes after 4 hour intervention on day1, day8, day16
  mood questionnaire(an abbreviated version of Profile of Mood States (POMS)) will be used before and after the intervention, such as tension, anger, depression, vigor, esteem-related effect, confusion, fatigue, total mood level data included. The scale is 0 to 4.
mood status assessed by confusion score | change from baseline all mood outcomes after 4 hour intervention on day1, day8, day16
  mood questionnaire(an abbreviated version of Profile of Mood States (POMS)) will be used before and after the intervention, such as tension, anger, depression, vigor, esteem-related effect, confusion, fatigue, total mood level data included. The scale is 0 to 4.
mood status assessed by fatigue score | change from baseline all mood outcomes after 4 hour intervention on day1, day8, day16
  mood questionnaire(an abbreviated version of Profile of Mood States (POMS)) will be used before and after the intervention, such as tension, anger, depression, vigor, esteem-related effect, confusion, fatigue, total mood level data included. The scale is 0 to 4.
mood status assessed by total mood level score | change from baseline all mood outcomes after 4 hour intervention on day1, day8, day16
  mood questionnaire(an abbreviated version of Profile of Mood States (POMS)) will be used before and after the intervention, such as tension, anger, depression, vigor, esteem-related effect, confusion, fatigue, total mood level data included. The scale is 0 to 4.
muscle activity | recording 5 minutes' muscle activity for each sitting posture, average RMS will be collected.it will be performed on another experiment day.
  Muscle activity is measured by the electromyograph （EMG）machine. RMS values will be collected and calculated as muscle activation during each sittings condition
discomfort level | report discomfort level immediately after each sitting condition(each sitting posture lasts 5 minutes).it will be performed on another experiment day.
  after each sitting condition, self discomfort level will be asked.0 means no discomfort,10 means the worst discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Hans HCM Savelberg, PhD, Study Director — Maastricht University
Locations (1):
- Faculty of Health, Medicine and Life Sciences, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
there is no sharing individual participant data